CLINICAL TRIAL: NCT02230306
Title: Phase II Study of Cobimetinib in Combination With Vemurafenib in Active Melanoma Brain Metastases
Acronym: CoBRIM-B
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: closed due to slow accrual
Sponsor: Melissa Burgess, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Melissa Burgess, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-123; ML29155 (Other: Genentech)
Record Dates: First submitted 2014-08-27; First posted 2014-09-03 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-09

CONDITIONS: Active Melanoma Brain Metastases
MeSH Terms: interventions — cobimetinib; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cobimetinib in Combination with Vemurafenib (Experimental): Vemurafenib (960 mg twice a day) will be taken on Days 1 - 28 of each 28-day treatment cycle. The first dose of vemurafenib should be taken in the morning, and the second dose should be taken in the evening. Vemurafenib can be taken with or without a meal and should be taken with a glass of water.
  Cobimetinib (60 mg once a day) will be taken on Days 1 - 21 of each 28-day treatment cycle. The cobimetinib tablet should be taken at approximately the same time each day in the morning with the vemurafenib dose, but no later than 4 hours after the scheduled time. Cobimetinib can be taken with or without a meal and should never be chewed, cut, or crushed and should be taken with a glass of water.
  Interventions: Drug: Cobimetinib; Drug: Vemurafenib

INTERVENTIONS:
Drug: Cobimetinib — 60mg once a day; will be taken on days 1-21 of each 28 day treatment cycle; will be taken in combination with Vemurafenib;
Drug: Vemurafenib — 960mg twice a day; 28 day treatment cycle; will be taken in combination with Cobimetinib;
  Other Names: Zelboraf

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the combination of vemurafenib with cobimetinib in patients with active melanoma brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically confirmed metastatic melanoma (Stage IV), carrying BRAF V600-mutation
* Melanoma must be documented to contain a BRAFV600 mutation by a CLIA approved laboratory
* At least one measurable intracranial target lesion for which all of the following criteria are met:

  1. previously untreated or progressive according to RECIST 1.1 (equal to or greater than 20% increase in longest diameter on baseline scan) after previous local therapy (SRS and/or craniotomy)
  2. immediate local therapy clinically not indicated or patient is not a suitable candidate to receive immediate local therapy (SRS and/or craniotomy)
  3. largest diameter of ≥ 0.5cm but ≤ 4 cm as determined by contrast-enhanced MRI
* Prior therapies for extracranial metastatic melanoma including chemo-, cytokine-, immuno-, biological- and vaccine-therapy will be allowed but prior BRAF or MEK not allowed
* ECOG PS 0-2
* Life expectancy >12 weeks
* Age 18 years or older
* Adequate bone marrow function as indicated by the following:

  1. ANC > 1500/µL
  2. Platelets ≥ 100,000/µL
  3. Hemoglobin > 9 g/dL
* Adequate renal function, as indicated by creatinine =/< 1.5 x the upper limit of normal (ULN)
* Adequate liver function, as indicated by bilirubin =/< 1.5 x ULN
* AST or ALT < 3 x ULN (patients with documented liver metastases: AST and/or ALT =/< 5 x ULN)
* Able to swallow pills
* Negative serum pregnancy test within 7 days prior to commencement of dosing in premenopausal women. Women of non-childbearing potential may be included without serum pregnancy test if they are either surgically sterile or have been postmenopausal for ≥ 1 year
* Fertile men and women must use an effective method of contraception during treatment and for at least 6 months after completion of treatment as directed by their physician. Effective methods of contraception are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (for example implants, injectables, combined oral contraception or intra-uterine devices). At the discretion of the Investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

* Active infection
* Prior therapy with BRAFi and/or MEKi
* Leptomeningeal disease
* Symptomatic brain metastases requiring immediate local interventions such as craniotomy or SRS
* Increasing corticosteroid dose in 7 days prior to administration of first dose of study drug. Symptomatic patients that have stable or decreasing corticosteroid use in the past 7 days will be allowed
* Current use of therapeutic warfarin
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI v4.0) [NCI, 2009] Grade 2 or higher from previous anti-cancer therapy, except alopecia
* Conditions that will interfere significantly with the absorption of drugs
* Inability to undergo MRI secondary to metal, claustrophobia, Gadolinium Contrast allergy
* Pregnant, lactating, or breast feeding women
* Prior radiation therapy within the last 14 days
* Concomitant malignancies or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Unwillingness or inability to comply with study and follow-up procedures
* The following foods/supplements are prohibited at least 7 days prior to initiation of and during study treatment:

  1. St. John's wort or hyperforin
  2. Grapefruit juice
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, Retinal Vein Occlusion (RVO), or neovascular macular degeneration
* Uncontrolled glaucoma with intra-ocular pressures > 21mmHg
* Serum cholesterol ≥ Grade 2
* Hypertriglyceridemia ≥ Grade 2
* Hyperglycemia (fasting) ≥ Grade 2
* History of clinically significant cardiac dysfunction, including the following:

  1. Current unstable angina
  2. Current symptomatic congestive heart failure of NYHA class 2 or higher
  3. History of congenital long QT syndrome or mean QTcF > 450 msec at baseline or uncorrectable electrolyte abnormalities
  4. Uncontrolled hypertension ≥ Grade 2 (patients with a history hypertension controlled with anti-hypertensives to ≤ Grade 1 are eligible)
  5. Left ventricular ejection fraction (LVEF) below 50%
  6. Uncontrolled Arrhythmias
  7. Myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack within the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Burgess, MD, Principal Investigator — University of Pittsburgh; Richard Carvajal, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Anna Pavlick, MD, Principal Investigator — NYU Clinical Cancer Center; Mohammed Milhem, MD, Principal Investigator — Univ of Iowa; Ravi Amaravadi, MD, Principal Investigator — Univ of Pennsylvania; Harriet Kluger, MD, Principal Investigator — Yale New Haven Hospital
Locations (6):
- United States (6):
  - Harriet Kluger, New Haven, Connecticut
  - Mohammed Milhem, MD, Iowa City, Iowa
  - Anna Pavlick, MD, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ravi Amaravadi, MD, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Cobimetinib in Combination With Vemurafenib: Vemurafenib (960 mg twice a day) taken on Days 1 - 28 of each 28-day treatment cycle. Cobimetinib (60 mg once a day) taken on Days 1 - 21 of each 28-day treatment cycle.
Period: Overall Study
Arm/Group | Cobimetinib in Combination With Vemurafenib
Started | 5
Completed | 4
Not Completed | 1
Not completed — Did not receive study treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cobimetinib in Combination With Vemurafenib
Number analyzed (Participants) | 5
Age, Customized [Number; unit: years]
  Patient 1 | 26
  Patient 2 | 65
  Patient 3 | 31
  Patient 4 | 33
  Patient 5 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Intracranial Response (OIRR)
Description: Change in overall size of the sum of diameters from baseline of up to 5 intracranial target lesions in response to study treatment, achieved by individual patients.
Time Frame: Until disease progression, less than or equal to 5 years.
Population: Patients who received study treatment and were assessed by MRI every 8 weeks.
Measure: Number; unit: centimeters
Arm/Group | Cobimetinib in Combination With Vemurafenib
Number analyzed (Participants) | 4
centimeters
  Patient #1 | -2.01
  Patient #2 | -0.8
  Patient #4 | -2.12
  Patient #5 | 0.6

2. Secondary Outcome: Overall Response
Description: Response to study treatment achieved by individual patients as indicated by an overall change in size of the sum of diameters from baseline of up to 5 intracranial target lesions and up to 5 extracranial target lesions.
Time Frame: Until disease progression, less than or equal to 5 years.
Population: Patients who received study treatment and were assessed by MRI every 8 weeks.
Measure: Number; unit: centimeters
Arm/Group | Cobimetinib in Combination With Vemurafenib
Number analyzed (Participants) | 4
centimeters
  Patient #1 | -6.61
  Patient #2 | -5.3
  Patient #4 | -9.12
  Patient #5 | -0.4

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Time (number of months) from first documented evidence of overall Complete Response (CR) or Partial Response (PR) until time of first documented disease progression or death due to any cause (for individual patients). Progression as defined by RECIST 1.1 (Response Evaluation Criteria In Solid Tumors) is a ≥ 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5mm.
Time Frame: Up to 5 years
Population: Patients who received study treatment and were assessed by MRI every 8 weeks.
Measure: Number; unit: months
Arm/Group | Cobimetinib in Combination With Vemurafenib
Number analyzed (Participants) | 4
months
  Patient #1 | 3.7
  Patient #2 | 3.7
  Patient #4 | 5.8
  Patient #5 | 1.7

4. Secondary Outcome: Overall Survival (OS)
Description: Number of months of survival for individual patients.
Time Frame: Up to 5 years
Measure: Number; unit: months
Arm/Group | Cobimetinib in Combination With Vemurafenib
Number analyzed (Participants) | 4
months
  Patient #1 | 7.3
  Patient #2 | 4.2
  Patient #4 | 5.8
  Patient #5 | 5.4

5. Secondary Outcome: Duration of Response
Description: Change in relative apparent diffusion coefficient (rADC) as measured by MRI as early predictor of response value/result for each patient
Time Frame: Until disease progression, less than or equal to 5 years.
Population: Patients for whom response duration data was obtainable in those that received MRI tumor assessments every 8 weeks.
Measure: Number; unit: months
Arm/Group | Cobimetinib in Combination With Vemurafenib
Number analyzed (Participants) | 3
months
  Patient #1 | 1.6
  Patient #2 | 1.8
  Patient #4 | 2.1

6. Secondary Outcome: Immune Modulation in Peripheral Blood
Time Frame: Up to 5 years
Population: Data were not able to be collected and thus zero participants were analyzed for this outcome.
Arm/Group | Cobimetinib in Combination With Vemurafenib
Number analyzed (Participants) | 0

7. Secondary Outcome: Early Markers of Progression in Peripheral Blood
Time Frame: Up to 5 years
Population: Zero participants were analyzed for this outcome.
Arm/Group | Cobimetinib in Combination With Vemurafenib
Number analyzed (Participants) | 0

8. Secondary Outcome: Health-related Quality of Life as Measured by The Functional Assessment of Cancer Therapy (FACT) - Brain (FACT-Br)
Description: The Functional Assessment of Cancer Therapy-Brain (FACT-Br) is used to measure general quality of life (QOL) that reflects symptoms or problems associated with brain malignancies across 5 scales. The brain subscale is usually used along with the core (general) questionnaire that includes 27 items. The measure yields information about total QOL, as well as information about the dimensions of physical well-being, social/family well-being, emotional well being, functional well-being, and disease-specific concerns. Patients rate all 5 items using a five-point Likert scale ranging from 0 "not at all" to 4 "very much." Overall, higher ratings suggest higher QOL. Items are totaled to produce the following subscales, along with an overall QOL score: physical well-being (7 items); social/family well-being (7 items); emotional well-being (6 items); functional well-being (7 items); and concerns relevant to patients with brain tumors (23 items). Scoring range is 0-200.
Time Frame: Up to 5 years
Measure: Number; unit: scores on a scale
Arm/Group | Cobimetinib in Combination With Vemurafenib
Number analyzed (Participants) | 4
scores on a scale
  Patient #1 - Cycle 1 | 107
  Patient #1 - Cycle 2 | 84
  Patient #1 - Cycle 3 | 110
  Patient #1 - Cycle 4 | 97
  Patient #2 - Cycle 1 | 83
  Patient #2 - Cycle 2 | 91
  Patient #2 - Cycle 3 | 104
  Patient #2 - Cycle 4 | 95
  Patient #4 - Cycle 1 | 98
  Patient #4 - Cycle 2 | 97
  Patient #4 - Cycle 3 | 95
  Patient #4 - Cycle 4 | 101
  Patient #4 - Cycle 5 | 119
  Patient #4 - Cycle 6 | 98
  Patient #5 - Cycle 1 | 69
  Patient #5 - Cycle 2 | 103
  Patient #5 - Cycle 3 | 104

ADVERSE EVENTS:
Arm/Group | Cobimetinib in Combination With Vemurafenib
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cobimetinib in Combination With Vemurafenib (N=4)
Papulopustular rash (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Neoplasms Benign, Malignant And Unspecified (Incl Cysts And Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hydrocephalus (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cobimetinib in Combination With Vemurafenib (N=4)
Anemia (Blood and lymphatic system disorders) | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 2
Photophobia (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Retinopathy (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Edema face (General disorders) | 1
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 3
Fever (General disorders) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
CPK increased (Investigations) | 2
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 2
GGT increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 4
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Lymphocyte count increased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Sinus pain (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes